CLINICAL TRIAL: NCT00834249
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Venlafaxine 25 mg Tablets and Effexor® 25 mg Tablets Administered as 1 x 25 mg Tablet in Healthy Subjects Under Fed Conditions
Brief Title: Venlafaxine 25 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 02355
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venlafaxine (Experimental): Venlafaxine 25 mg Tablet (test) dosed in first period followed by Effexor® 25 mg Tablet (reference) dosed in second period
  Interventions: Drug: Venlafaxine 25 mg Tablets
- Effexor® (Active Comparator): Effexor® 25 mg Tablet (reference) dosed in first period followed by Venlafaxine 25 mg Tablet (test) dosed in second period
  Interventions: Drug: Effexor® 25 mg Tablets

INTERVENTIONS:
Drug: Venlafaxine 25 mg Tablets — 1 x 25 mg, single-dose fasting
  Arms: Venlafaxine
Drug: Effexor® 25 mg Tablets — 1 x 25 mg, single-dose fasting
  Arms: Effexor®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of venlafaxine 25 mg tablets (test) versus Effexor® (reference) administered as 1 x 25 mg tablet under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females and/or males, non-smokers, 18 years of age and older. Female subjects will be post-menopausal or surgically sterilized.
* Post-menopausal status is defined as absence of menses for the past 12 months or hysterectomy with bilateral oophorectomy at least 6 months ago.
* Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks of the administration of study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90 mmHg; or heart rate less than 50 or over 100 bpm) at screening.
* Subjects with BMI ≥ 30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 Unit - 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* History of allergic reactions to venlafaxine.
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* History or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within the 90 days preceding study drug administration.
* Intolerance to venipuncture.
* Subjects with a clinically significant history of tuberculosis, epilepsy, asthma, diabetes, psychosis, or glaucoma will not be eligible for this study.
* Subjects who are unable to understand or unwilling to sign the Informed Consent Form.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical sub-investigator, contraindicates the subject's participation in this study.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 Days. Donation or loss of whole blood prior to administration of the study medication as follows: less than 300 mL of whole blood within 30 days or; 300 mL to 500 mL of whole blood within 45 days or; more than 500 mL of whole blood within 56 days.
* Subjects who have consumed food or beverages containing grapefruit (e.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.
* Subjects with known presence of volume-depletion.
* Subjects predisposed to bleeding of the skin and mucous membrane.
* Subjects with history or known presence of impaired platelet aggregation.
* Subjects with history of seizures.
* Breast-feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-12; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bicrell, M.D., Principal Investigator — Anapharm
Locations (2):
- Canada (2):
  - Anapharm Inc., Montreal, Quebec
  - Anapharm Inc., Sainte-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Venlafaxine (Test) First: Venlafaxine 25 mg Tablet (test) dosed in first period followed by Effexor® 25 mg Tablet (reference) dosed in second period
- Effexor® (Reference) First: Effexor® 25 mg Tablet (reference) dosed in first period followed by Venlafaxine 25 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Venlafaxine (Test) First | Effexor® (Reference) First
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Venlafaxine (Test) First | Effexor® (Reference) First
Started | 9 | 9
Completed | 8 | 8
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | Venlafaxine (Test) First | Effexor® (Reference) First
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venlafaxine (Test) First | Effexor® (Reference) First | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 8 | 9 | 17
  Black | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Venlafaxine in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Venlafaxine: Venlafaxine 25 mg Tablet (test) dosed in either period
- Effexor®: Effexor® 25 mg Tablet (reference) dosed in either period
Arm/Group | Venlafaxine | Effexor®
Number analyzed (Participants) | 15 | 15
ng/mL | 47.13 (18.19) | 46.45 (20.28)
Statistical Analysis 1: Comparison: Venlafaxine vs Effexor®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Test/Ref Ratio of LS Means x 100 = 101.73 — Bioequivalence is established when ratio of means falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated) - Venlafaxine in Plasma
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Venlafaxine | Effexor®
Number analyzed (Participants) | 15 | 15
ng*h/mL | 427.09 (357.42) | 422.70 (349.50)
Statistical Analysis 1: Comparison: Venlafaxine vs Effexor®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 99.73 — Bioequivalence is established when ratio of means falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant) - Venlafaxine in Plasma
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Venlafaxine | Effexor®
Number analyzed (Participants) | 15 | 15
ng*h/mL | 366.94 (255.01) | 366.50 (261.20)
Statistical Analysis 1: Comparison: Venlafaxine vs Effexor®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 99.71 — Bioequivalence is established when ratio of means falls within 80-125

4. Secondary Outcome: Cmax - O-Desmethylvenlafaxine in Plasma
Description: Informational Purposes Only
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Venlafaxine | Effexor®
Number analyzed (Participants) | 15 | 15
ng/mL | 75.15 (32.88) | 69.17 (31.46)
Statistical Analysis 1: Comparison: Venlafaxine vs Effexor®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 109.61 — Metabolite results not subjected to bioequivalence criteria, results are presented for informational purposes only

5. Secondary Outcome: AUC0-inf - O-desmethylvenlafazine in Plasma
Description: Informational Purposes Only
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Venlafaxine | Effexor®
Number analyzed (Participants) | 15 | 15
ng*h/mL | 1390.43 (555.40) | 1315.02 (552.49)
Statistical Analysis 1: Comparison: Venlafaxine vs Effexor®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 106.85 — Metabolite results not subjected to bioequivalence criteria, results are presented for informational puposes only

6. Secondary Outcome: AUC0-t - O-desmethylvenlafaxine in Plasma
Description: Informational Purposes Only
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Venlafaxine | Effexor®
Number analyzed (Participants) | 15 | 15
ng*h/mL | 1016.24 (425.24) | 960.47 (407.72)
Statistical Analysis 1: Comparison: Venlafaxine vs Effexor®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 106.38 — Metabolite results not subjected to bioequivalence criteria, results are presented for informational purposes only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.